CLINICAL TRIAL: NCT01369043
Title: Modulation of Insulin and Exercise Responses by Vitamin E and Vitamin C
Brief Title: The Effects of Vitamin E and Vitamin C and Exercise
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of successful recruiting, budget cuts, and potential study flaws.
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: GFHNRC503
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Exercise and Non-exercise Effect Upon Vitamins E and C
Keywords: Vitamin E; Vitamin C; Exercise; Antioxidant
MeSH Terms: conditions — Motor Activity | interventions — Vitamin E; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin E and Vitamin C (Active Comparator): 4 weeks with Vitamin E and Vitamin C supplementation with no exercise and 4 weeks of supplementation with prescribed exercise.
  Interventions: Dietary Supplement: Vitamin E and Vitamin C
- Placebo (No Intervention): Placebos instead of the Vitamin E and Vitamin C supplements

INTERVENTIONS:
Dietary Supplement: Vitamin E and Vitamin C — Vitamin E 400 iu/dose daily times 56 days Vitamin C 500 mg/dose twice daily times 56 days
  Arms: Vitamin E and Vitamin C

SUMMARY:
Moderate exercise is thought to be one of the best known means to improve how insulin works in people. Taking vitamin C and vitamin E is also thought to have the same effect. This study is being done to see if taking vitamin C and vitamin E improves or hinders how insulin works when people do not exercise and when they do exercise.

DETAILED DESCRIPTION:
The objective of the study is to determine in humans whether anti-oxidant supplementation with ascorbate (vitamin C) or R,R,R-α-tocopherol acetate (vitamin E) improves insulin sensitivity in the untrained state but blocks exercise-induced increases in insulin sensitivity and other adaptations to exercise. The results will provide new information on the roles of anti-oxidant supplementation in modifying insulin sensitivity, and will inform guidelines for anti-oxidant supplementation as an adjunct to exercise.

ELIGIBILITY:
Inclusion Criteria:

* 30 to 50 years of age
* Willing to not change eating habits
* Willing to not change physical activity habits
* Willing to complete the 28 week study
* Able to swallow pills

Exclusion Criteria:

* smoke or use tobacco or nicotine in any form including snuff, pills, and patches
* take any medication that makes you unable to do hard exercise
* have cardiovascular, pulmonary, and/or a metabolic disease such as diabetes
* have uncontrolled high blood pressure
* have alcohol, anabolic steroids, or other substance abuse issues
* consume more than 3 alcoholic drinks/week
* have any joint or muscle injuries that affects your ability to exercise
* have cancer (other than skin cancer or carcinoma in situ of the cervix)
* are pregnant or nursing

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
(1) Blood glucose and insulin following glucose challenge in non-exercising and exercising people (BMI 27 to 35) taking anti-oxidants (vitamin E and vitamin C) or placebo. | 28 weeks
  Individuals will be in placebo and vitamin supplemented groups in a cross-over design. A total of 6 oral glucose tolerance tests will be performed per subject in the study.

SECONDARY OUTCOMES:
(1) Resting metabolic rate, body composition, plasma oxidative stress, plasma vitamin E and vitamin C levels in non-exercising and exercising people (BMI 27 to 35) taking anti-oxidants (vitamin E and vitamin C) or placebo. | 28 weeks
(2) Fitness measures (heart rate, exercise work, VO2, VCO2, blood lactate) in non-exercising and exercising people (BMI 27 to 35) taking anti-oxidants (vitamin E and vitamin C) or placebo. | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Picklo, PhD, Principal Investigator — Agriculture Research Service, United States Department of Agriculture, Grand Forks Human Nutrition Research Center
Locations (1):
- Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

REFERENCES:
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Hathcock JN, Azzi A, Blumberg J, Bray T, Dickinson A, Frei B, Jialal I, Johnston CS, Kelly FJ, Kraemer K, Packer L, Parthasarathy S, Sies H, Traber MG. Vitamins E and C are safe across a broad range of intakes. Am J Clin Nutr. 2005 Apr;81(4):736-45. doi: 10.1093/ajcn/81.4.736. PMID 15817846
- [Background] Devaraj S, Leonard S, Traber MG, Jialal I. Gamma-tocopherol supplementation alone and in combination with alpha-tocopherol alters biomarkers of oxidative stress and inflammation in subjects with metabolic syndrome. Free Radic Biol Med. 2008 Mar 15;44(6):1203-8. doi: 10.1016/j.freeradbiomed.2007.12.018. Epub 2007 Dec 23. PMID 18191645
- [Background] Vincent HK, Bourguignon CM, Weltman AL, Vincent KR, Barrett E, Innes KE, Taylor AG. Effects of antioxidant supplementation on insulin sensitivity, endothelial adhesion molecules, and oxidative stress in normal-weight and overweight young adults. Metabolism. 2009 Feb;58(2):254-62. doi: 10.1016/j.metabol.2008.09.022. PMID 19154960
- [Background] Furukawa S, Fujita T, Shimabukuro M, Iwaki M, Yamada Y, Nakajima Y, Nakayama O, Makishima M, Matsuda M, Shimomura I. Increased oxidative stress in obesity and its impact on metabolic syndrome. J Clin Invest. 2004 Dec;114(12):1752-61. doi: 10.1172/JCI21625. PMID 15599400
- [Background] Gletsu-Miller N, Hansen JM, Jones DP, Go YM, Torres WE, Ziegler TR, Lin E. Loss of total and visceral adipose tissue mass predicts decreases in oxidative stress after weight-loss surgery. Obesity (Silver Spring). 2009 Mar;17(3):439-46. doi: 10.1038/oby.2008.542. Epub 2008 Dec 11. PMID 19219062
- [Background] Manning PJ, Sutherland WH, Walker RJ, de Jong SA, Berry EA. The effect of glucose ingestion on inflammation and oxidative stress in obese individuals. Metabolism. 2008 Oct;57(10):1345-9. doi: 10.1016/j.metabol.2008.04.020. PMID 18803936
- [Background] Manning PJ, Sutherland WH, Walker RJ, Williams SM, de Jong SA, Berry EA. The effect of rosiglitazone on oxidative stress and insulin resistance in overweight individuals. Diabetes Res Clin Pract. 2008 Aug;81(2):209-15. doi: 10.1016/j.diabres.2008.04.015. Epub 2008 Jun 9. PMID 18541328
- [Background] Sutherland WH, Manning PJ, Walker RJ, de Jong SA, Ryalls AR, Berry EA. Vitamin E supplementation and plasma 8-isoprostane and adiponectin in overweight subjects. Obesity (Silver Spring). 2007 Feb;15(2):386-91. doi: 10.1038/oby.2007.546. PMID 17299112
- [Background] Manning PJ, Sutherland WH, Walker RJ, Williams SM, De Jong SA, Ryalls AR, Berry EA. Effect of high-dose vitamin E on insulin resistance and associated parameters in overweight subjects. Diabetes Care. 2004 Sep;27(9):2166-71. doi: 10.2337/diacare.27.9.2166. PMID 15333479
- [Background] Perticone F, Ceravolo R, Candigliota M, Ventura G, Iacopino S, Sinopoli F, Mattioli PL. Obesity and body fat distribution induce endothelial dysfunction by oxidative stress: protective effect of vitamin C. Diabetes. 2001 Jan;50(1):159-65. doi: 10.2337/diabetes.50.1.159. PMID 11147782
- [Background] Chen H, Karne RJ, Hall G, Campia U, Panza JA, Cannon RO 3rd, Wang Y, Katz A, Levine M, Quon MJ. High-dose oral vitamin C partially replenishes vitamin C levels in patients with Type 2 diabetes and low vitamin C levels but does not improve endothelial dysfunction or insulin resistance. Am J Physiol Heart Circ Physiol. 2006 Jan;290(1):H137-45. doi: 10.1152/ajpheart.00768.2005. Epub 2005 Aug 26. PMID 16126809
- [Background] Rizzo MR, Abbatecola AM, Barbieri M, Vietri MT, Cioffi M, Grella R, Molinari A, Forsey R, Powell J, Paolisso G. Evidence for anti-inflammatory effects of combined administration of vitamin E and C in older persons with impaired fasting glucose: impact on insulin action. J Am Coll Nutr. 2008 Aug;27(4):505-11. doi: 10.1080/07315724.2008.10719732. PMID 18978171
- [Background] Bailey DM, Davies B, Young IS, Jackson MJ, Davison GW, Isaacson R, Richardson RS. EPR spectroscopic detection of free radical outflow from an isolated muscle bed in exercising humans. J Appl Physiol (1985). 2003 May;94(5):1714-8. doi: 10.1152/japplphysiol.01024.2002. Epub 2003 Mar 7. PMID 12626489
- [Background] Bailey DM, Lawrenson L, McEneny J, Young IS, James PE, Jackson SK, Henry RR, Mathieu-Costello O, McCord JM, Richardson RS. Electron paramagnetic spectroscopic evidence of exercise-induced free radical accumulation in human skeletal muscle. Free Radic Res. 2007 Feb;41(2):182-90. doi: 10.1080/10715760601028867. PMID 17364944
- [Background] Bailey DM, Young IS, McEneny J, Lawrenson L, Kim J, Barden J, Richardson RS. Regulation of free radical outflow from an isolated muscle bed in exercising humans. Am J Physiol Heart Circ Physiol. 2004 Oct;287(4):H1689-99. doi: 10.1152/ajpheart.00148.2004. Epub 2004 May 20. PMID 15155256
- [Background] Mastaloudis A, Leonard SW, Traber MG. Oxidative stress in athletes during extreme endurance exercise. Free Radic Biol Med. 2001 Oct 1;31(7):911-22. doi: 10.1016/s0891-5849(01)00667-0. PMID 11585710
- [Background] Mastaloudis A, Morrow JD, Hopkins DW, Devaraj S, Traber MG. Antioxidant supplementation prevents exercise-induced lipid peroxidation, but not inflammation, in ultramarathon runners. Free Radic Biol Med. 2004 May 15;36(10):1329-41. doi: 10.1016/j.freeradbiomed.2004.02.069. PMID 15110397
- [Background] Mastaloudis A, Traber MG, Carstensen K, Widrick JJ. Antioxidants did not prevent muscle damage in response to an ultramarathon run. Med Sci Sports Exerc. 2006 Jan;38(1):72-80. doi: 10.1249/01.mss.0000188579.36272.f6. PMID 16394956
- [Background] Mastaloudis A, Yu TW, O'Donnell RP, Frei B, Dashwood RH, Traber MG. Endurance exercise results in DNA damage as detected by the comet assay. Free Radic Biol Med. 2004 Apr 15;36(8):966-75. doi: 10.1016/j.freeradbiomed.2004.01.012. PMID 15059637
- [Background] Ristow M, Zarse K, Oberbach A, Kloting N, Birringer M, Kiehntopf M, Stumvoll M, Kahn CR, Bluher M. Antioxidants prevent health-promoting effects of physical exercise in humans. Proc Natl Acad Sci U S A. 2009 May 26;106(21):8665-70. doi: 10.1073/pnas.0903485106. Epub 2009 May 11. PMID 19433800
- [Background] Gomez-Cabrera MC, Domenech E, Romagnoli M, Arduini A, Borras C, Pallardo FV, Sastre J, Vina J. Oral administration of vitamin C decreases muscle mitochondrial biogenesis and hampers training-induced adaptations in endurance performance. Am J Clin Nutr. 2008 Jan;87(1):142-9. doi: 10.1093/ajcn/87.1.142. PMID 18175748